CLINICAL TRIAL: NCT01227928
Title: A Study to Evaluate Efficacy and Safety of Pazopanib Monotherapy in Asian Women Who Have Not Progressed After First-line Chemotherapy for Advanced Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma - An Extension Study to VEG110655
Brief Title: Efficacy and Safety of Pazopanib Monotherapy After First-line Chemotherapy in Ovarian, Fallopian Tube, or Primary Peritoneal Cancer in Asian Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114012
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms, Ovarian
Keywords: tyrosine kinase inhibitors; Primary Peritoneal Carcinoma; primary peritoneal cancer; ovarian cancer; Fallopian Tube Cancer; gynecologic cancer; anti-angiogenesis; pazopanib
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pazopanib (Experimental): experimental medication
  Interventions: Drug: Pazopanib
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800 mg daily for 24 months
  Arms: pazopanib
Drug: Placebo comparator — Placebo 800 mg daily for 24 months
  Arms: placebo

SUMMARY:
This is a study to determine whether therapy with pazopanib is effective and safe in Asian women with epithelial ovarian, fallopian tube or primary peritoneal cancer whose cancer has not progressed on first-line chemotherapy.

DETAILED DESCRIPTION:
This study is an extension study to the VEG110655 study. The parent study, VEG110655, was designed to evaluate whether pazopanib 800 mg daily for 52 weeks will prolong progression free survival (PFS) in women diagnosed with ovarian, fallopian tube or primary peritoneal cancer. These women will have obtained stable disease, a complete remission, or a partial remission after debulking surgery and at least five cycles of chemotherapy (taxane/platinum). This extension study will evaluate safety and efficacy outcomes of pazopanib monotherapy and placebo in an Asian population with the same indication as the parent study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* At least 18 years old.
* Histologically confirmed, International Federation of Gynecology and Obstetrics (FIGO) stage II-IV epithelial ovarian, fallopian tube or primary peritoneal carcinoma that was treated with surgical debulking and at least five cycles of platinum-taxane doublet chemotherapy.
* Study randomization at least 3 weeks and not more than 12 weeks from the date of the last chemotherapy dose, and all major toxicities from the previous chemotherapy must have resolved.
* No evidence of disease progression
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Able to swallow and retain oral medication.
* Adequate hematologic, hepatic, and renal system function as follows:

Hematologic

* Absolute neutrophil count (ANC) at least 1.5 X 10^9/L
* Hemoglobin at least 9 g/dL (or 5.59 mmol/L)
* Platelets at least 100 X 10^9/L
* Prothrombin time (PT) or international normalized ratio (INR) up to 1.2 X ULN
* Activated partial thromboplastin time (aPTT) up to 1.2 X ULN Hepatic
* Total bilirubin up to 1.5 X ULN
* AST and ALT up to 2.5 X ULN Renal
* Serum creatinine up to 1.5 mg/dL

Or, if greater than 1.5 mg/dL:

Calculated creatinine clearance at least 50 mL/min Urine Protein

* Urine protein is 0, trace, or +1 determined by dipstick urinalysis, or < 1.0 gram determined by 24-hour urine protein analysis.
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) OR childbearing potential, and agrees to use adequate contraception.

Exclusion Criteria:

* Either (a) bulky disease, or (b) any residual disease which in the opinion of the investigator will need imminent second-line therapy
* Synchronous primary endometrial carcinoma, or a past history of primary endometrial carcinoma, are excluded unless certain conditions are met.
* Clinically significant gastrointestinal abnormalities
* Prolongation of corrected QT interval (QTc) > 480 msecs
* History of any one or more cardiovascular conditions within the past 6 months prior to randomization
* Poorly controlled hypertension
* History of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months prior to randomization
* Major surgery (including interval debulking) or trauma within 28 days, or minor surgical procedures within 7 days, prior to randomization, or has any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Hemoptysis within 6 weeks prior to randomization.
* Endobronchial metastases.
* Serious and/or unstable pre-existing medical (e.g., uncontrolled infection), psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Investigational or anti-VEGF anticancer therapy prior to study randomization.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.
* Prior or concurrent invasive malignancies that currently or within the last 5 years show/ed activity of disease (except ovarian, fallopian tube, or peritoneal cancer, or concurrent endometrial cancer FIGO stages IA/B)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- China (8):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Hong Kong, Hong Kong
- GSK Investigational Site, Seoul, South Korea
- GSK Investigational Site, Taipei, Taiwan

REFERENCES:
- [Derived] Kim JW, Mahner S, Wu LY, Shoji T, Kim BG, Zhu JQ, Takano T, Park SY, Kong BH, Wu Q, Wang KL, Ngan HY, Liu JH, Wei LH, Mitrica I, Zhang P, Crescenzo R, Wang Q, Cox CJ, Harter P, du Bois A. Pazopanib Maintenance Therapy in East Asian Women With Advanced Epithelial Ovarian Cancer: Results From AGO-OVAR16 and an East Asian Study. Int J Gynecol Cancer. 2018 Jan;28(1):2-10. doi: 10.1097/IGC.0000000000000602. PMID 26588236

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching placebo administered orally once daily for up to 24 months.
- Pazopanib 800 Milligrams: Participants received pazopanib 800 milligrams administered orally once daily for up to 24 months.
Period: Overall Study
Arm/Group | Placebo | Pazopanib 800 Milligrams
Started | 72 | 73
Completed | 50 | 56
Not Completed | 22 | 17
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pazopanib 800 Milligrams | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (10.46) | 51.7 (9.62) | 52.9 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 73 | 145
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time interval between randomization and evidence of progressive disease (PD), as assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, or death, whichever occurred first. A visit-based analysis approach to determine participants' dates of progression was applied in the analysis method. PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Participants who were alive and had not progressed at the time of analysis were censored at the date associated with the last visit with adequate assessment.
Time Frame: From randomization until evidence of progressive disease or death, whichever occurred first (average of 15.2 months)
Population: Intent-to-Treat (ITT) Population: all randomized participants who were not screen failures. Participants who were screen failures and randomized by mistake, but who did not receive study treatment, were not included. The treatment assignment in the ITT Population was based on the randomized treatment. The data cut off was October 12, 2012.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 73
months | 18.1 [12.1 to NA] — The lower and upper bounds of the confidence intervals were calculated when there was a sufficient number of events (progressions or deaths). | 18.1 [18.0 to 18.1]
Statistical Analysis 1: Comparison: Placebo vs Pazopanib 800 Milligrams; Test type: Superiority or Other; Hazard Ratio (HR) = 0.984, 95% CI 2-sided [0.595 to 1.626] — The Hazard Ratio (HR) is estimated using a Pike estimator. The HR was adjusted for the stratification factor of first-line treatment outcome

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time interval from the date of randomization to the date of death due to any cause.
Time Frame: From randomization until death due to any cause (average of 29.4 months)
Population: ITT Population. Participants who were alive as of study completion were censored at the last contact date. The cut off for these data was January 10, 2014.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 73
months | NA [NA to NA] — There were too few events of death for median overall survival or the 95% confidence interval to be reached. | NA [NA to NA] — There were too few events of death for median overall survival or the 95% confidence interval to be reached.
Statistical Analysis 1: Comparison: Placebo vs Pazopanib 800 Milligrams; Test type: Superiority or Other; p = 0.5901, Log Rank; Hazard Ratio (HR) = 0.811, 95% CI 2-sided [0.376 to 1.751] — The Hazard Ratio (HR) is estimated using a Pike estimator. The HR was adjusted for the three stratification factors

3. Secondary Outcome: PFS by Gynaecologic Cancer Intergroup (GCIG) Criteria
Description: PFS by GCIG criteria is defined as the time from the randomization date to the earliest date of disease progression (PD) per GCIG criteria or death due to any cause. Per GCIG criteria, an objective progression is defined as the earliest event of either tumor progression based on RECIST v1.0 or confirmed CA-125 progression. A participant is counted as "Progressed per RECIST" if the radiological PD per RECIST occurred prior to or on the same day as CA-125 progression. A participant is counted as "Progressed per CA-125" if the radiological PD occurred after CA-125 progression. Per RECIST, PD is defined as at least a 20% increase in the sum of the LD of target lesions, taking as a reference, the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Participants who were alive and had not progressed at the time of analysis were censored at the date associated with the last visit with adequate assessment.
Time Frame: From randomization to the earliest date of disease progression per GCIG criteria or death due to any cause (average of 15.2 months)
Population: ITT Population. The cut off for these data was October 12, 2012.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 73
months | 15.2 [9.0 to NA] — The lower and upper bounds of the confidence intervals were calculated when there was a sufficient number of events (progressions or deaths). | 16.1 [14.2 to 18.2]

4. Secondary Outcome: Number of Participants With Any Dose Reduction or Any Dose Interruption
Description: Dose interruptions or reductions may have been required following potential drug-related toxicities. As a general rule, if dose reduction of investigational product (IP) was necessary, the dose should have been reduced stepwise by 200 mg at each step, and the participant should have been monitored for 10 to 14 days. If toxicity recurred or worsened during this monitoring time, the IP could have been interrupted and/or the dose of IP further decreased, with continued monitoring for an additional 10 to 14 days, and so on. The cut off for these data was October 12, 2012.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population: all randomized participants who received at least one dose of investigational product. Treatment assignments in the All Treated Population were based on the actual treatment received, if different from the randomized treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Any Reduction | 26 | 64
  Any Interruption | 44 | 65

5. Secondary Outcome: Number of Participants With Any Non-serious Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalizaton or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. See the non-serious AE/SAE module for a list of specific events.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population: all randomized participants who received at least one dose of investigational product. Treatment assignments in the All Treated Population were based on the actual treatment received, if different from the randomized treatment. The cut off for these data was January 10, 2014.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Any AE | 65 | 72
  Any SAE | 4 | 7

6. Secondary Outcome: Number of Participants With Any On-therapy AE and Any AE Related to Study Treatment
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. On-therapy AEs were those reported from the first day that randomized study drug was received to 28 days after the last dose of randomized study drug, and within 28 days of dose interruption. Relatedness was assessed by the Investigator.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Any on-therapy AE | 65 | 72
  Any AE related to study treatment | 52 | 71

7. Secondary Outcome: Number of Participants With Any Grade 3 or 4 AE
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. The NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0 was used to grade AEs per the following scale to assess severity: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling AE; Grade 5, death related to AE.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants | 8 | 39

8. Secondary Outcome: Number of Participants With the Indicated On-therapy Grade 3-5 AEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. On-therapy AEs were those reported from the first day that randomized study drug was received to 28 days after the last dose of randomized study drug, and within 28 days of dose interruption. The NCI-CTCAE Version 3.0 was used to grade AEs per the following scale to assess severity: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling AE; Grade 5, death related to AE. ALT=alanine aminotransferase; AST=aspartate aminotransferase.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Hypertension, Grade 3 | 1 | 13
  Neutropenia, Grade 3 | 0 | 9
  Leukopenia, Grade 3 | 0 | 1
  Diarrhea, Grade 3 | 1 | 5
  ALT increased, Grade 3 | 0 | 1
  Thrombocytopenia, Grade 3 | 0 | 3
  AST increased, Grade 3 | 0 | 1
  Neutrophil count decreased, Grade 3 | 0 | 2
  Neutrophil count decreased, Grade 4 | 0 | 1
  Arthralgia, Grade 3 | 0 | 1
  Upper respiratory tract infection, Grade 3 | 1 | 0
  Protein urine, Grade 3 | 0 | 1
  Proteinuria, Grade 3 | 0 | 1
  Bone pain, Grade 3 | 0 | 1
  Toothache, Grade 3 | 0 | 1
  Pyrexia, Grade 3 | 1 | 0
  Hepatic function abnormal, Grade 3 | 0 | 1
  Liver injury, Grade 3 | 0 | 1
  Abdominal distension, Grade 3 | 1 | 0
  Bradycardia, Grade 3 | 0 | 1
  Febrile neutropenia, Grade 3 | 0 | 1
  Thrombus in device, Grade 3 | 0 | 1
  Pruritis, Grade 3 | 1 | 0
  Amylase increased, Grade 3 | 1 | 0
  Cerebral ischaemia, Grade 3 | 1 | 0
  Foot fracture, Grade 3 | 1 | 0

9. Secondary Outcome: Number of Participants With AEs Leading to Permanent Discontinuation of Study Treatment, Dose Interruption, and Dose Reduction
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Dose interruptions or reductions may have been required following potential drug-related toxicities. As a general rule, if dose reduction of investigational product (IP) was necessary, the dose should have been reduced stepwise by 200 mg at each step, and the participant should have been monitored for 10 to 14 days. If toxicity recurred or worsened during this monitoring time, the IP could have been interrupted and/or the dose of IP further decreased, with continued monitoring for an additional 10 to 14 days, and so on.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Permanent discontinuation | 1 | 18
  Dose interruption | 29 | 67
  Dose reduction | 24 | 63

10. Secondary Outcome: Number of Participants With Any SAE, Any SAE Related to Study Treatment, and Any Fatal SAE
Description: An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalizaton or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. See the non-serious AE/SAE module for a list of specific events. Relatedness was assessed by the Investigator.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Any SAE | 4 | 7
  Any SAE related to study treatment | 1 | 4
  Any fatal SAE | 0 | 0

11. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Blood Pressure Shifts From Baseline
Description: Systolic blood pressure (SBP) and Diatolic blood pressure (DBP) are measured in millimeters of mercury (mmHg). A participant could have been counted in more than one shift category. Participants who experienced shifts in both SBP and DBP are represented under each individual parameter. A worst-case on-therapy shift is defined as the worst shift that occurred at any time during the treatment period.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population. One participant on placebo did not report any blood pressure measurements post-Baseline. The cut off for these data was January 10, 2014.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 71 | 72
participants
  SBP, Any increase to >=120 mmHg | 28 | 53
  SBP, Increase to 140-<160 mmHg | 4 | 23
  SBP, Increase to >=160 mmHg | 0 | 6
  DBP, Any increase to >=80 mmHg | 35 | 59
  DBP, Increase to 90-<100 mmHg | 1 | 25
  DBP, Increase to >=100 mmHg | 0 | 5

12. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Shift From Baseline in Bazett's Corrected QT Interval (QTc)
Description: 12-lead ECGs were obtained at the scheduled visits. A worst-case on-therapy shift is defined as the worst shift that occurred at any time during the treatment period. The QTc is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. In general, the faster the heart rate the shorter the QTc. If a QTc >=500 milliseconds (msec) was noted on a scheduled or unscheduled electrocardiogram (ECG), then two additional ECGs should have been obtained within 5 minutes to confirm the abnormality. The average QTc was determined from the three ECG tracings by manual evaluation and was used to determine continued eligibility.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population. Only those participants for which a post-Baseline ECG was conducted were analyzed. The cut off for these data was October 12, 2012.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 69 | 70
participants
  Any increase to >=450 msec | 10 | 5
  Increase to 481-500 msec | 1 | 1
  Increase to >=501 msec | 2 | 0

13. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Hematology Parameter Grade Shifts From Baseline Grade
Description: Grade shifts from Baseline were assessed as any grade increase (AGI), increase to Grade (G) 3 (ITG3), and increase to Grade 4 (ITG4). Toxicities were graded according to the National Cancer Institute common toxicity criteria (NCI-Common Toxicity Criteria for Adverse Events), version 4.0. Grade refers to the severity of the toxicity. The CTCAE displays Grades (G) 1 through 5 with unique clinical descriptions of severity for each toxicity based on the following general guideline: G1, mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; G2, moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); G3, severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; G4, Life-threatening consequences; urgent intervention indicated.; G5, death related to AE.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population. Data are presented for only those participants with laboratory values. The cut off for these data was October 12, 2012.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 69 | 71
participants
  Hemoglobin, AGI | 4 | 14
  Hemoglobin, ITG3 | 0 | 0
  Hemoglobin, ITG4 | 0 | 0
  Lymphocytes, AGI | 11 | 9
  Lymphocytes, ITG3 | 2 | 1
  Lymphocytes, ITG4 | 0 | 0
  Neutrophils, AGI | 22 | 55
  Neutrophils, ITG3 | 0 | 11
  Neutrophils, ITG4 | 0 | 2
  Platelets, AGI | 10 | 32
  Platelets, ITG3 | 0 | 1
  Platelets, ITG4 | 0 | 0
  White blood cells, AGI | 19 | 48
  White blood cells, ITG3 | 0 | 2
  White blood cells, ITG4 | 0 | 0

14. Secondary Outcome: Number of Participants With the Indicated Worst-case On-therapy Chemistry Parameter Grade Shifts From Baseline Grade
Description: as for outcome 13
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 69 | 70
participants
  Albumin, AGI, n=69, 70 | 2 | 1
  Albumin, ITG3, n=69, 70 | 0 | 0
  Albumin, ITG4, n=69, 70 | 0 | 0
  Creatinine, AGI, n=69, 70 | 2 | 2
  Creatinine, ITG3, n=69, 70 | 0 | 1
  Creatinine, ITG4, n=69, 70 | 0 | 0
  Hypercalcemia, AGI, n=69, 69 | 9 | 3
  Hypercalcemia, ITG3, n=69, 69 | 1 | 0
  Hypercalcemia, ITG4, n=69, 69 | 0 | 0
  Hyperglycemia, AGI, n=69, 70 | 16 | 14
  Hyperglycemia, ITG3, n=69, 70 | 0 | 0
  Hyperglycemia, ITG4, n=69, 70 | 0 | 0
  Hyperkalemia, AGI, n=69, 70 | 0 | 1
  Hyperkalemia, ITG3, n=69, 70 | 0 | 0
  Hyperkalemia, ITG4, n=69, 70 | 0 | 0
  Hypermagnesemia, AGI, n=69, 69 | 6 | 2
  Hypermagnesemia, ITG3, n=69, 69 | 1 | 1
  Hypermagnesemia, ITG4, n=69, 69 | 0 | 0
  Hypernatremia, AGI, n=69, 70 | 2 | 3
  Hypernatremia, ITG3, n=69, 70 | 0 | 0
  Hypernatremia, ITG4, n=69, 70 | 0 | 0
  Hypocalcemia, AGI, n=69, 69 | 4 | 5
  Hypocalcemia, ITG3, n=69, 69 | 0 | 0
  Hypocalcemia, ITG4, n=69, 69 | 0 | 0
  Hypoglycemia, AGI, n=69, 70 | 0 | 3
  Hypoglycemia, ITG3, n=69, 70 | 0 | 0
  Hypoglycemia, ITG4, n=69, 70 | 0 | 0
  Hypokalemia, AGI, n=69, 70 | 10 | 6
  Hypokalemia, ITG3, n=69, 70 | 0 | 0
  Hypokalemia, ITG4, n=69, 70 | 0 | 0
  Hypomagnesemia, AGI, n=69, 69 | 6 | 2
  Hypomagnesemia, ITG3, n=69, 69 | 0 | 0
  Hypomagnesemia, ITG4, n=69, 69 | 0 | 0
  Hyponatremia, AGI, n=69, 70 | 1 | 1
  Hyponatremia, ITG3, n=69, 70 | 0 | 0
  Hyponatremia, ITG4, n=69, 70 | 0 | 0
  Phosphate, AGI, n=69, 69 | 2 | 4
  Phosphate, ITG3, n=69, 69 | 0 | 0
  Phosphate, ITG4, n=69, 69 | 0 | 0

15. Secondary Outcome: Number of Participants With the Indicated Worst-case Eastern Cooperative Oncology Group (ECOG) Performance Status Shifts From Baseline Grades of 0, 1, and 2
Description: The ECOG performance status scales and criteria are used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. Grade 5, dead.
Time Frame: From Week 1 until the end of the treatment period (up to Study Week 108)
Population: All Treated Population. The cut off for these data was October 12, 2012.
Measure: Number; unit: participants
Arm/Group | Placebo | Pazopanib 800 Milligrams
Number analyzed (Participants) | 72 | 72
participants
  Baseline score of 0; shift to 0 | 56 | 46
  Baseline score of 0; shift to 1 | 2 | 13
  Baseline score of 0; shift to 2 | 0 | 0
  Baseline score of 1; shift to 0 | 0 | 0
  Baseline score of 1; shift to 1 | 12 | 13
  Baseline score of 1; shift to 2 | 1 | 0
  Baseline score of 2; shift to 0 | 0 | 0
  Baseline score of 2; shift to 1 | 0 | 0
  Baseline score of 2; shift to 2 | 1 | 0

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the All Treated Population, comprised of all randomized participants who received at least one dose of investigational product. Treatment assignments in the All Treated Population were based on the actual treatment received, if different from the randomized treatment.
Arm/Group | Placebo | Pazopanib 800 Milligrams
Serious Adverse Events (participants affected / at risk) | 4/72 | 7/72
Other Adverse Events (participants affected / at risk) | 59/72 | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Pazopanib 800 Milligrams (N=72)
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Cerebral artery stenosis (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Pazopanib 800 Milligrams (N=72)
Hypertension (Vascular disorders) | 20 | 55
Neutropenia (Blood and lymphatic system disorders) | 16 | 46
Leukopenia (Blood and lymphatic system disorders) | 18 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 17
Diarrhoea (Gastrointestinal disorders) | 5 | 35
Abdominal pain (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 3 | 11
Abdominal pain upper (Gastrointestinal disorders) | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 29
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 21
Rash (Skin and subcutaneous tissue disorders) | 8 | 4
Alanine aminotransferase increased (Investigations) | 4 | 19
Aspartate aminotransferase increased (Investigations) | 6 | 16
Blood thyroid stimulating hormone increased (Investigations) | 2 | 15
Blood lactate dehydrogenase increased (Investigations) | 2 | 7
Neutrophil count decreased (Investigations) | 2 | 6
Blood bilirubin increased (Investigations) | 1 | 5
Protein urine present (Investigations) | 1 | 6
Electrocardiogram QT prolonged (Investigations) | 4 | 0
Headache (Nervous system disorders) | 5 | 13
Dizziness (Nervous system disorders) | 3 | 10
Nasopharyngitis (Infections and infestations) | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Urinary tract infection (Infections and infestations) | 6 | 5
Fatigue (General disorders) | 8 | 14
Chest discomfort (General disorders) | 3 | 4
Pyrexia (General disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 8
Proteinuria (Renal and urinary disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.